CLINICAL TRIAL: NCT03088293
Title: A Multicenter Randomized Open-label Trial Comparing the Efficacy and Safety of Infliximab Versus Cyclophosphamide in Subjects With Idiopathic Refractory Scleritis
Brief Title: Cyclophosphamide vs. Infliximab for Refractory Idiopathic Scleritis (CIRIS)
Acronym: CIRIS
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: recruiting difficulties
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL17_0028; 2017-004969-27 (EudraCT Number)
Record Dates: First submitted 2017-03-17; First posted 2017-03-23 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Idiopathic Refractory Scleritis
Keywords: idiopathic refractory scleritis; infliximab; cyclophosphamide
MeSH Terms: interventions — Infliximab; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- infliximab (Experimental): Patients will receive prednisone and infliximab (5 mg/kg at week 0, 2, 6, 11 and 16 as an intravenous (IV) infusion) in association with low-dose methotrexate (10 mg/week) for 16 weeks.
  Interventions: Drug: Infliximab
- cyclophosphamide (Experimental): Patients will receive prednisone and cyclophosphamide intravenously (700 mg/m2 every 4 weeks intravenously) (n=25) for 16 weeks.
  Interventions: Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Infliximab — Patients will receive prednisone and infliximab (5 mg/kg at week 0, 2, 6, 11 and 16 as an intravenous (IV) infusion) in association with low-dose methotrexate (10 mg/week) for 16 weeks.
  Arms: infliximab
Drug: Cyclophosphamide — Patients will receive prednisone and cyclophosphamide intravenously (700 mg/m2 every 4 weeks intravenously) (n=25) for 16 weeks.
  Arms: cyclophosphamide

SUMMARY:
This study will evaluate the Efficacy and Safety of Infliximab versus Cyclophosphamide in Subjects with Idiopathic Refractory Scleritis.

The term scleritis describes a chronic inflammation that involves the outermost cost and skeleton of the eye. Scleritis is classified anatomically as either anterior or posterior based on the principal location of the inflammation. Thirty to forty percent of scleritis cases are associated with systemic autoimmune conditions including rheumatoid arthritis and granulomatosis with polyangiitis. Infectious causes including herpes virus and varicella zoster account for 5 to 10% of patients. The remaining 50% of cases are classified as idiopathic.

CIRIS, is the first prospective randomized, head to head study, comparing infliximab to cyclophosphamide in refractory idiopathic scleritis. There is no firm evidence or randomized controlled trials directly addressing the best biologic agent in severe and refractory idiopathic scleritis. If left untreated or insufficiently treated, scleritis can progress to peripheral ulcerative keratitis, uveitis and glaucoma. Visual loss occurs in approximately 10% of patients with anterior scleritis and in up to 75% of patients with posterior scleritis. The incidence of burden in ocular inflammation (uveitis and scleritis) has been dramatically reduced in the recent years with the use of biologics, raising the question of whether these compounds should be used earlier in the treatment of severe non infectious scleritis. Contrasting with other immunosuppressors, cyclophosphamide and infliximab act rapidly and are highly effective in steroid's sparing.

Despite a strong rationale, these compounds are not yet approved in idiopathic refractory scleritis, which guarantees the innovative nature of this study that aims selecting or dropping any arm when evidence of efficacy already exists.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to the performance of any study-specific procedures
2. Male or female, subject aged > or = 18 at Screening
3. Weight 40 - 120 kg at Screening
4. Diagnosis of anterior idiopathic scleritis or anterior and posterior idiopathic scleritis at least one eye. Scleritis is classified anatomically as anterior based on the principal location of the inflammation. Clinically, anterior scleritis can be divided into diffuse, nodular or necrotizing types.
5. Active disease: Currently uncontrolled scleritis disease. Uncontrolled scleritis disease is defined as (at least) a 2 in sclera inflammation, according to the grading system defined by Sene for sclera inflammation (gradings from 0 to 4).
6. Refractory disease: At screening, subjects must be receiving oral corticosteroids (>10 mg/day prednisone equivalent and <80 mg/day) and at least one other immunosuppressive for more than 4 months (azathioprine, methotrexate, mycophenolate mofetyl, cyclosporine, leflunomide) or be intolerant to such immunosuppressive therapies.
7. Topical corticosteroids and/or NSAIDs are permitted provided the dose regimen has been stable for 2 weeks prior to Screening and remains stable throughout the study. Topical treatment for cycloplegia is permitted.

   Page 40 sur 129
8. Chest X-ray results (postero-anterior and lateral) within 12 weeks prior to the randomization visit with no evidence of active Tuberculosis, active infection, or malignancy.
9. For female subjects of child-bearing age, a negative serum pregnancy test. A woman is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient (definition of the Clinical Trial Facilitation Group).
10. For subjects with reproductive potential, a willingness to use adequate contraceptive measures to prevent the subject or the subject's partner from becoming pregnant during the study. For women in period of childbearing adequate contraceptive measures include hormonal methods used for two or more cycles prior to Screening and 6 months after the last dose treatment should be used (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly, or condom used in conjunction with contraceptive foam or jelly), intrauterine devices (IUD), sterilization (e.g., tubal ligation or a monogamous relationship with a vasectomized partner), and abstinence. For men who are sexually active with a women in period of childbearing adequate contraceptive measures from screening to 6 months after the last dose treatment should be used (For men: barrier methods (condom used in conjunction with contraceptive foam or jelly), sterilization (vasectomy) and abstinence. For his partner: hormonal methods (e.g., oral contraceptive pills, contraceptive patch, or contraceptive vaginal ring), barrier methods (e.g., contraceptive sponge, diaphragm used in conjunction with contraceptive foam or jelly), intrauterine devices (IUD), sterilization (e.g., tubal ligation)).
11. A negative QuantiFERON®-Tuberculosis (TB) test result or, in the event that their QuantiFERON®-TB test result at Screening is positive, all subjects must agree to complete an INH treatment course of at least 6 months.
12. Affiliated to the French social security system.

Exclusion Criteria:

1. medical contraindication to administer experimental drugs: Cyclophosphamide (urinary obstruction, bladder inflammation…) or Infliximab (moderate or severe heart failure, classe III /IV classification NYHA…)/low dose Methotrexate (chronic respiratory insufficiency…); and non-experimental drugs (10 % phenylephrine instillation, prednisone, paracetamol, polaramine, folic acid and uromitexan)
2. Infectious scleritis, posterior idiopathic scleritis or scleritis related to systemic diseases (i.e. granulomatosis with polyangiitis, rheumatoid arthritis, lupus, relapsing chondritis, etc)
3. Blindness or very low visual acuity (<1/20) of the no study eye
4. Active tuberculosis or history of untreated tuberculosis
5. Known positive syphilis serology, HIV antibody, . Positive serology for hepatitis B or C virus is not considered as non-inclusion criteria. These tests should be performed during the screening, and in case of positive result the opinion of a hepatologist will be requested
6. History of malignancy within 5 years prior to Screening other than carcinoma in situ of the cervix or adequately treated, non-metastatic squamous or basal cell carcinoma of the skin.
7. History of severe allergic or anaphylactic reactions to monoclonal antibodies. Hypersensitivity known to cyclophosphamide, to infliximab, to other murine proteins, to methotrexate or to any of the excipients.
8. Infectious disease:

   1. Fever or infection requiring treatment with antibiotics within 3 weeks prior to Screening or between Screening and Day 0.
   2. History of recurrent infection or predisposition to infection.
9. Known immunodeficiency
10. History of multiple sclerosis and/or demyelinating disorder
11. Laboratory values assessed during Screening:

    1. Hemoglobin <8.5 g/dL
    2. WBC <3.0 x 103/mm3
    3. Platelet count <100 x 103/mm3
    4. Glomerular filtration rates (GFR) <30 ml/min.
    5. AST/ALT >1.5 x upper limit of normal (ULN)
    6. Absolute Neutrophil Count <2.0 x 103/mm3
    7. Absolute Lymphocyte Count <0.5 x 103/mm3
12. Use of the following systemic treatments during the specified periods:

    1. Any other previous systemic biological therapy, including anti-TNF
    2. Treatment with any systemic alkylating agents within 12 months prior to Screening or between Screening and Day 0 (e.g., cyclophosphamide, chlorambucil)
    3. Any live (attenuated) vaccine within 3 months prior to Screening or between Screening and Day 0; recombinant or killed virus vaccines are permitted. Live seasonal flu and H1N1 vaccines are permitted ≥2 weeks prior to Screening.
13. Participation to another interventional research.
14. Inability to understand information concerning the protocol.
15. Pregnant or lactating women.
16. Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-11 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with resolution (score=0) of the scleral inflammation and with a prednisone dose lower than 0.1 mg/kg/day | Week 20
  Scleritis will be graded and scored according to the grading system defined by Sen for sclera inflammation (gradings from 0 to 4): these findings will be documented by drawings, photography or both for central review.

SECONDARY OUTCOMES:
percentage of patients with a decrease of at least 2 in sclera inflammation with a prednisone dose lower or equal to 0.1 mg/kg/day. | Week 20
  according to Sen and al gradation at week 20 and with a prednisone dose lower or equal to 0.1 mg/kg/day.
Mean change in sclera inflammation from baseline to Week 20. | Week 20
  from baseline to Week 20 (according to Sen and al gradation)
Time to response onset (total resolution in sclera inflammation). | Week 26
Mean change in Best corrected visual acuity | Week 20
  from baseline to week 20 (ETDRS letter score)
percentage of patients meeting targets: ≤ 0.1 mg/day prednisone | Week 20
mean change dose of corticosteroid | Week 26
  * mean dose at week 20,
  * cumulative dose.
Mean dose of corticosteroid | Week 20
Cumulative dose of corticosteroid | Week 26
Frequency to relapse of scleritis | Week 26
  Relapse will be diagnosed when inflammation will restart within 6 months of tapering or discontinuation of medication.Early relapse will be distinguished to later relapse. Early relapse corresponds to any scleritis relapse within the 3 months after discontinuation of medication and later relapse corresponds to any scleritis relapse after 3 months after discontinuation of medication.
Characteristics of scleritis at worsening. | Week 26
Frequency to relapse of scleritis and the characteristics of scleritis at worsening. | Week 52
  Relapse will be diagnosed when inflammation will restart within 6 months of tapering or discontinuation of medication.Early relapse will be distinguished to later relapse. Early relapse corresponds to any scleritis relapse within the 3 months after discontinuation of medication and later relapse corresponds to any scleritis relapse after 3 months after discontinuation of medication.
Characteristics of scleritis at worsening. | Week 52
Time to relapse of scleritis | Week 26
  Relapse will be diagnosed when inflammation will restart within 6 months of tapering or discontinuation of medication. Early relapse will be distinguished to later relapse. Early relapse corresponds to any scleritis relapse within the 3 months after discontinuation of medication and later relapse corresponds to any scleritis relapse after 3 months after discontinuation of medication.
Time to relapse of scleritis | Week 52
  Relapse will be diagnosed when inflammation will restart within 6 months of tapering or discontinuation of medication. Early relapse will be distinguished to later relapse. Early relapse corresponds to any scleritis relapse within the 3 months after discontinuation of medication and later relapse corresponds to any scleritis relapse after 3 months after discontinuation of medication.
Mean change in quality of life | Week 16 ; Week 26
  assessed using the 36-Item Short Form Health Survey (SF-36) - from baseline to W16 and W26
Mean change in of vision-related quality of life | Week 16 ; Week 26
  assessed by the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) - from baseline to W16 and W26

CONTACTS AND LOCATIONS:
Overall Officials: Pascal SEVE, Principal Investigator — Hospices Civils de Lyon - Hopital de la Croix Rousse - Médecine Interne